CLINICAL TRIAL: NCT06241924
Title: Oscillatory Activity in Basal Ganglia Circuits During Normal and Pathological Movement
Acronym: BAG-OSMOV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CHUBX 2022/80
Record Dates: First submitted 2024-01-26; First posted 2024-02-05 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Parkinson Disease; Epilepsy
Keywords: Focal seizure; Parkinson disease; Hyperkinetic seizures; Hypokinetic disorders; Dyskinesia; Networks; Basal ganglia
MeSH Terms: conditions — Parkinson Disease; Epilepsy; Seizures; Dyskinesias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epilepsy (Experimental)
  Interventions: Procedure: Stereo-electro-encephalography (SEEG)
- parkinson disease (Experimental)
  Interventions: Procedure: High Resolution Electroencephalogram (EEG-HR)

INTERVENTIONS:
Procedure: High Resolution Electroencephalogram (EEG-HR) — Local field potentials (LFP) recording using EEG-HR
  Arms: parkinson disease
Procedure: Stereo-electro-encephalography (SEEG) — Local field potentials (LFP) recording using sEEG
  Arms: Epilepsy

SUMMARY:
The expression of hypokinetic and hyperkinetic motor symptoms is accompanied by pathological synchronous oscillations of neuronal activity in this cortico-subcortical network with a wide frequency range.

The purpose of this research is to study cortico-subcortical oscillations and their synchronization in two pathologies emblematic of hypokinetic (Parkinson's disease) and hyperkinetic (epilepsies) phenomena using a simple motor task and comparing different situations.

DETAILED DESCRIPTION:
In order to define the link between the characteristics of the oscillations (frequency, amplitude, phase relation) within this cortico-subcortical network and movement (normal or pathological) in humans, a simple motor task of gripping/pulling a lever has been designed.

The local field potentials (LFPs) will be collected during the same motor task in :

i) patients with Parkinson's disease, using a high-resolution electroencephalogram (EEG) and the PERCEPT(TM) system (Medtronic) equipped with a "sensing" function for deep LFP recordings and in EEG-HR (for high resolution) for cortical recordings

ii) patients with focal drug-resistant epilepsy, during a pre-surgical assessment by stereo-electro-encephalography (SEEG). The SEEG allows the recording of both the cortex and the subcortical regions in a concomitant manner, and a direct correlation can be studied.

ELIGIBILITY:
Inclusion criteria :

* Male or Female
* Between 18 and 75 years of age
* With Parkinson's disease and already operated with implantation of electrodes in the Subthalamic nucleus connected to a PERCEPT (TM) device.
* Giving free, informed, written consent signed by the participant and the investigator Or
* With drug-resistant epilepsy and benefiting from a phase II pre-surgical assessment with intracerebral electrophysiological exploration by stereo-EEG
* With at least one electrode exploring the basal ganglia or the thalamus.
* Able to perform the simple motor task
* Affiliated or beneficiary of a social security scheme;
* Giving free, informed, written consent signed by the participant and the investigator

Exclusion criteria:

* Be incapable of giving consent personally
* Be subject to a legal protection measure or be placed under judicial protection;
* Being pregnant or breastfeeding
* Present a serious and/or decompensated somatic or psychiatric illness

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2027-02-05 (Estimated); Study Completion 2027-02-05 (Estimated)

PRIMARY OUTCOMES:
difference in the cortico-subcortical electrophysiological coherence value | Day 1
  difference in the cortico-subcortical electrophysiological coherence value between normal movement (control condition) and hypo- or hyperkinetic pathological movement

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme AUPY, Docteur, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France